CLINICAL TRIAL: NCT06166927
Title: The Correlation Between Ultrasound-measured Styloid Process of the Distal Radius and the Outer Diameter of the Best-fitting Endotracheal Tube in Pediatrics
Brief Title: The Use of a US-measured Styloid Process of the Distal Radius EET Diameter for Prediction of ETT Size
Acronym: ETT/US
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar. MD, Professor, Assiut University
Other Study IDs: 04-2023-200515
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Airway Management
Keywords: Children, airway, ETT, US, radial diameter

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cuffed Endotracheal tube.: Patients will be intubated using a high-volume low-pressure cuffed ETT with its OD determined by US measurement of the epiphyseal diameter of the distal radius.
  Interventions: Device: Cuffed endotracheal tube
- Uncuffed Endotracheal tube.: Patients will be intubated using an uncuffed ETT with its OD determined by US measurement of the epiphyseal diameter of the distal radius.
  Interventions: Device: UnCuffed ETT

INTERVENTIONS:
Device: Cuffed endotracheal tube — Patients will be intubated using a cuffed ETT with its OD determined by US measurement of the epiphyseal diameter of the distal radius.
  Other Names: Cuffed ETT
  Groups: Cuffed Endotracheal tube.
Device: UnCuffed ETT — Patients will be intubated using an uncuffed ETT (Flexicare-UK) with its OD determined by US measurement of the epiphyseal diameter of the distal radius.
  Other Names: Patients will be intubated using an uncuffed ETT with its OD determined by US measurement of the epiphyseal diameter of the distal radius.
  Groups: Uncuffed Endotracheal tube.

SUMMARY:
This study will aim to test the accuracy of the ultrasonography measurement of the epiphyseal diameter of the distal radius in the prediction of the size of the cuffed and uncuffed ETT that best fits in children (1-6 years old) in comparison with the traditional age-based formulas.

DETAILED DESCRIPTION:
Various formulas are used to predict the inner diameter (ID) of the ETT tube whether uncuffed or cuffed based on weight, age, height, and finger size. The accuracy of these formulas is questionable. These formulas depend on the child's demographic characteristics assuming that he/she has normal growth and development and cannot be applied to children with altered growth and development. Moreover, these formulas predict the ID of the ETT ignoring the tube thickness and the OD of the selected tube.

ultrasound has recently been identified as an accurate alternative to these formulas. The US-measured epiphyseal diameter of the distal radius is a method that has been recently introduced as a surrogate for the tracheal diameter. The issue is that the size of the airway can be considered a reflection of the body's growth, assuming that the growth rates of the cartilage all over the body are closely related to each other. Therefore, the measurement of the growth of the bony cartilage of the hand can be considered a surrogate marker of the tracheal diameter.9 The extent to which ultrasonography by this method can succeed in predicting the optimal pediatric ETT size remains under investigation.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 10-30 kg.
* Age: 1-6 years.
* Sex: both males and females.
* ASA physical status: I-II.
* Operation: elective surgery in which airway management with an endotracheal tube is needed.

Exclusion Criteria:

* Upper airway malformations.
* Upper airway surgery.
* Active respiratory illness (cough, fever, rhinorrhea) on the day of anesthesia,
* Anticipated difficult airway.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 1-6 years of both sexes undergoing surgical procedures in which an endotracheal tube is needed.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Agreement between the reference tube size based on US- Epiphyseal Diameter of distal radius measured OD and the final BFT | At induction of anesthesia
  The US probe will be first placed longitudinally over the distal radius to identify the epiphysis. Then the probe will be turned 90 degrees to identify and measure the transverse diameter of the radius epiphysis. These measured diameters coincide with the OD of the ETT.

CONTACTS AND LOCATIONS:
Overall Officials: Hala S Abdel-Ghaffar, MD, Principal Investigator — Assiut University
Locations (1):
- Assiut university Pediatric hospital, Asyut, Assiut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No